CLINICAL TRIAL: NCT07154355
Title: Clinical Study Protocol on the Impact of Community-Based Exercise Training on the Exercise Capacity of Patients With Reduced Cardiovascular and Pulmonary Function
Brief Title: Community Exercise Treating Effect on Cardiopulmonary Disease Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-148
Record Dates: First submitted 2025-01-25; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-01

CONDITIONS: Coronary Heart Disease (CHD); Heart Failure; Cardiomyopathy; COPD; Bronchial Asthma; Respiratory Failure; Thoracic Tumors; Cardiopulmonary Diseases
MeSH Terms: conditions — Coronary Disease; Heart Failure; Cardiomyopathies; Pulmonary Disease, Chronic Obstructive; Asthma; Respiratory Insufficiency; Pulmonary Heart Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- community-based exercise group (Experimental)
- non-exercise group (No Intervention)

INTERVENTIONS:
Behavioral: community-based exercise training — The patients will engage in 40-60 minutes of exercise training, either at home or in the community, five times a week, for eight weeks. Brisk walking, jogging, swimming, cycling, and trekking were among the exercise modalities that were chosen mostly based on the patient's individual preferences and habits. To guarantee safe and efficient exercise, exercise intensity was modified based on each person's subjective effort level and the results of their individual cardiorespiratory exercise tests.

SUMMARY:
The goal of this clinical trial is to learn if community-based exercise training can benefit patients aged 18 to 85 with diminished cardiovascular and pulmonary function. The main aim of this study is:

• Establish a community or home-based fitness training program for patients with cardiopulmonary insufficiency to improve adherence, safety, and efficacy while alleviating the burden on both patients and society.

Researchers will compare community-based exercise training to non-exercise training to see if community-based exercise training works to improve cardiovascular and pulmonary function.

Participants will:

* Engage in community or home exercise training for 40-60 minutes, five times weekly, during a duration of eight weeks. Exercise modalities are primarily determined by the patients' individual preferences and habits, such as brisk walking, running, swimming, cycling, and hiking.
* Adjust the exercise intensity according to their cardiopulmonary exercise test and the person's perceived exertion level.
* Utilize fitness bracelets or watches to document statistics during workouts and submit them to the experimenter weekly, covering the five days of exercise within that week.
* refrain from making any dietary modifications throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 85 with abnormal pulmonary or cardiovascular function.
2. Individuals who have completed a medical screening form to confirm they are free from illnesses and prescription medications that could impair their ability to complete the required testing and fitness training.
3. Participants who did not engage in structured, systematic moderate-to-intense strength or endurance training during the study period (specifically, not within the previous year).
4. At the onset of the trial, participants were physically active but had never participated in formal exercise more than twice a week.

Exclusion Criteria:

1. Patients with neuromuscular or skeletal disorders, or systemic diseases such as diabetes, cancer, or heart disease.
2. Individuals using medications known to affect health or the interpretation of study results.
3. Participants who have engaged in organized, systematic endurance or strength training of moderate to high intensity within the past year.
4. Patients who decline to participate in the study.
5. Other medical conditions or states that render exercise training inappropriate.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
exercise capacity | at enrollment and week 8
  Peak oxygen uptake (peakVO₂, ml/(kg·min)), measured by cardiopulmonary exercise testing (CPET), refers to the maximum rate of oxygen consumption per unit time during exhaustive incremental exercise. It serves as a key indicator of cardiopulmonary function and aerobic metabolic capacity.
exercise capacity | at enrollment and week 8
  Anaerobic Threshold (AT, mmol/L) is a key physiological parameter in cardiopulmonary exercise testing (CPET), representing the transition point from predominantly aerobic to anaerobic metabolism during incremental exercise. It is determined by measuring blood lactate concentration through serial blood sampling and plotting the lactate-exercise intensity curve.
life quality | at enrollment and week 8
  The Short Form-36 Health Survey (SF-36) was administered, with scores ranging from 0 to 100 across its eight subscales. Higher scores reflect superior health-related quality of life (HRQoL).

SECONDARY OUTCOMES:
Other exercise capacity outcome | at enrollment and week 8
  Exercise time
Other exercise capacity outcome | at enrollment and week 8
  The 6-minute walk distance (6MWD, m) , obtained through the 6-minute walk test (6MWT), refers to the maximum distance a patient can walk at their fastest pace on a flat, hard surface within 6 minutes. It is used to evaluate an individual's functional exercise capacity and cardiopulmonary endurance.
Other exercise capacity outcome | at enrollment and week 8
  Ventilatory anaerobic threshold (VAT, mL/(kg·min)) , a key physiological parameter in cardiopulmonary exercise testing (CPET), is determined by synchronously monitoring ventilatory parameters during incremental exercise (treadmill/cycle ergometer) and plotting the ventilation-intensity curve. It marks the transition point from predominantly aerobic to anaerobic metabolism during graded exercise.
Other exercise capacity outcome | at enrollment and week 8
  Ventilation/carbon dioxide (VE/VCO₂, mL/(kg·min)) slope, a key parameter for assessing ventilatory efficiency in cardiopulmonary exercise testing (CPET), is defined as the linear regression slope of minute ventilation (VE) against carbon dioxide output (VCO₂), reflecting the volume of ventilation required to eliminate 1 liter of CO₂ during exercise.
Leg strength | at enrollment and week 8
  The Nottingham strength test device is used to assess lower limb muscle strength, with a focus on measuring leg extensor power. By calculating the ratio of power output to body weight (power/weight), it indirectly reflects muscle functional status.
cardiac function | at enrollment and week 8
  Left ventricular ejection fraction (LVEF, %), measured by Doppler echocardiography, is used to assess left ventricular systolic function, representing the percentage of blood pumped out per heartbeat relative to the left ventricular end-diastolic volume.
Blood indices | at enrollment and week 8
  B-type natriuretic peptide (BNP, pg/mL), a key biomarker for heart failure, is used in the diagnosis and therapeutic monitoring of cardiovascular diseases such as heart failure.
Blood indices | at enrollment and week 8
  High-sensitivity C-reactive protein (hsCRP, mg/L) , an inflammatory biomarker measured by high-sensitivity detection technology, is used for cardiovascular disease risk assessment, infection monitoring, and chronic inflammation evaluation.
Blood indices | at enrollment and week 8
  Plasma interleukin-6 (IL-6, pg/mL) levels, a multifunctional proinflammatory cytokine, are used to assess systemic inflammation levels

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation Medicine Guangdong Provincial People's Hospital (Guangdong Academy of Medical Sciences), Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Hawley-Hague H, Horne M, Campbell M, Demack S, Skelton DA, Todd C. Multiple levels of influence on older adults' attendance and adherence to community exercise classes. Gerontologist. 2014 Aug;54(4):599-610. doi: 10.1093/geront/gnt075. Epub 2013 Jul 30. PMID 23899623
- [Background] Farrance C, Tsofliou F, Clark C. Adherence to community based group exercise interventions for older people: A mixed-methods systematic review. Prev Med. 2016 Jun;87:155-166. doi: 10.1016/j.ypmed.2016.02.037. Epub 2016 Feb 24. PMID 26921655
- [Background] Salmon P. Effects of physical exercise on anxiety, depression, and sensitivity to stress: a unifying theory. Clin Psychol Rev. 2001 Feb;21(1):33-61. doi: 10.1016/s0272-7358(99)00032-x. PMID 11148895
- [Background] Bashi N, Karunanithi M, Fatehi F, Ding H, Walters D. Remote Monitoring of Patients With Heart Failure: An Overview of Systematic Reviews. J Med Internet Res. 2017 Jan 20;19(1):e18. doi: 10.2196/jmir.6571. PMID 28108430
- [Background] Peek K, Sanson-Fisher R, Mackenzie L, Carey M. Interventions to aid patient adherence to physiotherapist prescribed self-management strategies: a systematic review. Physiotherapy. 2016 Jun;102(2):127-35. doi: 10.1016/j.physio.2015.10.003. Epub 2015 Oct 22. PMID 26821954
- [Background] Boggenpoel BY, Nel S, Hanekom S. The use of periodized exercise prescription in rehabilitation: a systematic scoping review of literature. Clin Rehabil. 2018 Sep;32(9):1235-1248. doi: 10.1177/0269215518769445. Epub 2018 Apr 17. PMID 29663831
- [Background] Jack K, McLean SM, Moffett JK, Gardiner E. Barriers to treatment adherence in physiotherapy outpatient clinics: a systematic review. Man Ther. 2010 Jun;15(3):220-8. doi: 10.1016/j.math.2009.12.004. Epub 2010 Feb 16. PMID 20163979
- [Background] O'Regan A, Pollock M, D'Sa S, Niranjan V. ABC of prescribing exercise as medicine: a narrative review of the experiences of general practitioners and patients. BMJ Open Sport Exerc Med. 2021 Jun 2;7(2):e001050. doi: 10.1136/bmjsem-2021-001050. eCollection 2021. PMID 34150320
- [Background] Oja P. Dose response between total volume of physical activity and health and fitness. Med Sci Sports Exerc. 2001 Jun;33(6 Suppl):S428-37; discussion S452-3. doi: 10.1097/00005768-200106001-00011. PMID 11427767
- [Background] Jakicic JM, Davis KK. Obesity and physical activity. Psychiatr Clin North Am. 2011 Dec;34(4):829-40. doi: 10.1016/j.psc.2011.08.009. Epub 2011 Oct 15. PMID 22098807
- [Background] Kehat I, Molkentin JD. Molecular pathways underlying cardiac remodeling during pathophysiological stimulation. Circulation. 2010 Dec 21;122(25):2727-35. doi: 10.1161/CIRCULATIONAHA.110.942268. No abstract available. PMID 21173361
- [Background] Kandola AA, Osborn DPJ, Stubbs B, Choi KW, Hayes JF. Individual and combined associations between cardiorespiratory fitness and grip strength with common mental disorders: a prospective cohort study in the UK Biobank. BMC Med. 2020 Nov 11;18(1):303. doi: 10.1186/s12916-020-01782-9. PMID 33172457
- [Background] Morkane CM, Kearney O, Bruce DA, Melikian CN, Martin DS. An Outpatient Hospital-based Exercise Training Program for Patients With Cirrhotic Liver Disease Awaiting Transplantation: A Feasibility Trial. Transplantation. 2020 Jan;104(1):97-103. doi: 10.1097/TP.0000000000002803. PMID 31205265
- [Background] Tutor A, Lavie CJ, Kachur S, Dinshaw H, Milani RV. Impact of cardiorespiratory fitness on outcomes in cardiac rehabilitation. Prog Cardiovasc Dis. 2022 Jan-Feb;70:2-7. doi: 10.1016/j.pcad.2021.11.001. Epub 2021 Nov 12. PMID 34780726
- [Background] Schmid D, Leitzmann MF. Cardiorespiratory fitness as predictor of cancer mortality: a systematic review and meta-analysis. Ann Oncol. 2015 Feb;26(2):272-8. doi: 10.1093/annonc/mdu250. Epub 2014 Jul 9. PMID 25009011
- [Background] Kodama S, Saito K, Tanaka S, Maki M, Yachi Y, Asumi M, Sugawara A, Totsuka K, Shimano H, Ohashi Y, Yamada N, Sone H. Cardiorespiratory fitness as a quantitative predictor of all-cause mortality and cardiovascular events in healthy men and women: a meta-analysis. JAMA. 2009 May 20;301(19):2024-35. doi: 10.1001/jama.2009.681. PMID 19454641
- [Background] Pedersen BK, Saltin B. Exercise as medicine - evidence for prescribing exercise as therapy in 26 different chronic diseases. Scand J Med Sci Sports. 2015 Dec;25 Suppl 3:1-72. doi: 10.1111/sms.12581. PMID 26606383
- [Background] Powell TA, Mysliwiec V, Brock MS, Morris MJ. OSA and cardiorespiratory fitness: a review. J Clin Sleep Med. 2022 Jan 1;18(1):279-288. doi: 10.5664/jcsm.9628. PMID 34437054
- [Background] Ferrari AU, Radaelli A, Centola M. Invited review: aging and the cardiovascular system. J Appl Physiol (1985). 2003 Dec;95(6):2591-7. doi: 10.1152/japplphysiol.00601.2003. PMID 14600164
- [Background] Zhou M, Wang H, Zeng X, Yin P, Zhu J, Chen W, Li X, Wang L, Wang L, Liu Y, Liu J, Zhang M, Qi J, Yu S, Afshin A, Gakidou E, Glenn S, Krish VS, Miller-Petrie MK, Mountjoy-Venning WC, Mullany EC, Redford SB, Liu H, Naghavi M, Hay SI, Wang L, Murray CJL, Liang X. Mortality, morbidity, and risk factors in China and its provinces, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2019 Sep 28;394(10204):1145-1158. doi: 10.1016/S0140-6736(19)30427-1. Epub 2019 Jun 24. PMID 31248666